CLINICAL TRIAL: NCT06518421
Title: The Role of Limbic Subcortical Structures and Cognition in Chronic Neuropathic Pain
Brief Title: Emotion and Memory in Chronic Neuropathic Pain
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Mojgan Hodaie, Senior Scientist, University Health Network, Toronto
Other Study IDs: 14-7350
Record Dates: First submitted 2024-03-01; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Trigeminal Neuralgia; Facial Pain
Keywords: Trigeminal Neuralgia; Facial Pain; Emotion; Cognition; Memory
MeSH Terms: conditions — Trigeminal Neuralgia; Facial Pain | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Controls: Brain imaging, clinical data, and cognitive data will be prospectively collect and analyze in both healthy control and patients with trigeminal neuralgia groups. Prospective data collection for control group includes:
  * MRI scan (1 timepoint)
  * Neuropsychological assessments (1 timepoint)
  Interventions: Behavioral: Neuropsychological assessments; Diagnostic Test: MR Imaging
- Trigeminal Neuralgia: Trigeminal Neuralgia is the most common chronic neuropathic facial pain disorder, characterized by the sudden onset of intermittent, intense, shock-like pain in distributions of the trigeminal nerve branches. TN has several unique features that distinguish it as an ideal model for the study of chronic pain: TN is largely unilateral; is severe in its nature; has stereotypical presentation among patients; and is not associated with other sensory deficits observed in other chronic pain disorders, such as numbness.
  Brain imaging, clinical data, and cognitive data will be prospectively collect and analyze in both healthy control and patients with trigeminal neuralgia groups. Prospective data collection for TN group includes:
  * MRI scan (2 timepoints; pre- and 6-month post-surgery)
  * Neuropsychological assessments (2 timepoints; pre- and 6-month post-surgery)
  Interventions: Behavioral: Neuropsychological assessments; Diagnostic Test: MR Imaging

INTERVENTIONS:
Behavioral: Neuropsychological assessments — * Pain questionnaires such as Numerical Pain Rating Scale is one of the most widely used multidimensional pain scales to assesses a person's pain based on the words they use to describe their pain.
  * Battery of Cognitive questionnaires = The cognitive test battery was designed to assess key cognitive abilities including attention, concentration, verbal learning and memory, verbal fluency, working memory and executive function as well as global cognitive functioning and fear and anxiety
  * Mnemonic Simulation Test and Rey Auditory Verbal Learning Test are the neuropsychological assessments designed to evaluate recognition and verbal memory, respectively. Both tasks have been shown to be very sensitive to hippocampal engagement and damage.
  * Memory-recall interview is an interview for the interviewees to recall the event from different perspectives, such as from the preadmission date, 2-week post- and 6-month post-surgical date. This supports the memory retrieval process.
Diagnostic Test: MR Imaging — Magnetic Resonance Imaging is a noninvasive medical imaging test that produces detailed images of almost every internal structure in the human body, including the organs, bones, muscles and blood vessels. MRI scanners create images of the body using a large magnet and radio waves.

SUMMARY:
Chronic pain affects one in four Canadians, leading to severe personal and societal costs. Over 70% of chronic pain patients report memory difficulties and fear having unexpected pain. Abnormalities in brain structures associated with emotion and memory, including the hippocampus and amygdala, can be affected by chronic pain. Understanding the relationship between chronic pain, structural brain changes, and cognitive functioning will lead to improved diagnosis, treatment, and outcomes in chronic pain disorders. In this project, the investigators will use advanced brain imaging techniques that assess the structure and function of the brain along with cognitive assessments to examine the overlap between chronic pain and emotion-memory processes. The study team will conduct the study using an excellent model of chronic pain-trigeminal neuralgia, a severe form of facial pain that responds well to surgical treatment. Brain images and cognitive data will be collected from participants before and after surgical treatment for pain. This information will be analyzed and compared with age- and sex-matched healthy individuals. This study will be the first to thoroughly investigate relationships between brain structure and function, cognition (memory, emotion), and promises to impact our understanding of chronic neuropathic pain conditions.

DETAILED DESCRIPTION:
Chronic pain affects 1 in 4 Canadians leading to severe personal and societal consequences. Over 70% of patients with chronic pain report cognitive deficits including memory difficulties and fear of having unexpected pain. However, the impact of chronic pain on cognition has not been adequately studied. Trigeminal neuralgia (TN), a severe facial pain with clear surgical outcomes, is an ideal model to address this question. Limbic structures, including the hippocampus (HPC) and amygdala (AMG), link emotion-memory and pain. Our prior CIHR-funded research revealed significant HPC volume reduction that normalized with successful treatment and abnormal HPC activity and AMG volume in chronic pain. These findings provide the foundation for a better understanding of the limbic subcortical structures and neuronal mechanisms of chronic pain.

Multimodal neuroimaging techniques have emerged as important tools for studying brain abnormalities in TN - seeking to elucidate the underlying neural mechanisms of HPC and AMG alterations, along with emotion-memory processes. This will be the first comprehensive study of limbic subcortical structural alterations and cognition in chronic pain.

Goal(s)/Research Aims

Our overall goal is to uncover the underlying neural mechanism of HPC and AMG alteration in TN and how these relate to chronic pain pathophysiology and cognition. Our specific aims are:

1. To characterize abnormalities in HPC subfields and their associated link with memory-specific performance in TN patients and their potential resolution following surgery.
2. To investigate the role of the AMG in pain-related fear in TN patients pre- and post-surgery and their associated link with the treatment outcomes.
3. To determine the relationship between the alterations in HPC subfields and the amygdaloid complex, and emotion-memory processes in TN patients pre- and post-surgery.

Methods/Approaches/Expertise The investigators will prospectively analyze brain imaging, clinical, and cognitive data from 340 participants (170 TN and 170 healthy age-/sex-matched controls). Patients will be scanned and assessed pre- and 6 months post-surgical treatment for TN.

In Aim 1, HPC subfield volumes will be extracted to characterize regional abnormalities in TN patients. The investigators will use HPC-sensitive memory tasks, including the mnemonic similarity task and the Rey Auditory Verbal Learning Test , to explore whether the HPC-specific memory processes correlate with structural abnormalities outlined.

In Aim 2, AMG nuclei volumes will be extracted to characterize regional abnormalities in TN patients. Fear of pain questionnaires and the Pain Catastrophizing Scale will be used to explore the link between pain-related fear and chronic pain.

In Aim 3, a validated fMRI task designed for episodic simulation based on novel word-pain associations will be used to examine the relationship between the abnormalities in the HPC subfields and AMG nuclei, and emotion-memory processes in TN patients pre- and post-surgery.

The NPA is a neurosurgeon and scientist with a strong clinical research focus on chronic pain. The team has expertise in chronic pain, brain imaging, cognition, and multivariate statistics.

Expected Outcomes Our innovative proposal interfaces brain imaging with cognition. Knowledge of the relationships between limbic structures, cognition, and pain will revolutionize pain assessment and treatment decisions. Uncovering neural mechanisms of HPC- and AMG-related structures in pain may improve healthcare delivery and patient outcomes by providing objective insights complementing current clinical care.

ELIGIBILITY:
Inclusion Criteria (for HC and TN):

* Age between 35 and 60 years old
* Absence of other active major neurological or psychiatric disorders
* Absence of MRI contraindications
* Able to communicate sufficiently to complete tasks and questionnaires
* Montreal Cognitive Assessment (MoCA) score greater than 23/30 (MoCA ≤23/30 could indicate severe cognitive impairment)

Inclusion Criteria for TN:

* Experiencing TN pain over a period of 6 months
* Stable medication use
* Meet established diagnostic criteria for TN (ICHD-3)

Exclusion Criteria (both HC and TN):

* Presence of other chronic pain/headache conditions
* Untreated hypertension or diabetes mellitus
* History of chronic drug or substance use disorder, chronic use of opioids or steroids, head trauma affecting cognitive performance,
* History/presence of active psychiatric illness and/or current use of psychoactive medication
* History of multiple sclerosis, skull base injury or tumours

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All gender identify including in Male, Female, Intersex, Bisexual, Asexual/Allies, Lesbian, Gay, Transgender/Transexual, Queer/Questioning, Cisgender, Non-binary, Genderqueer, Two-spirit, and Gender neutral are welcome to participate in this study.
Study Population: * Healthy control will be recruited from the local community
  * Patients with Trigeminal neuralgia will be recruited through our Neurosurgery and Pain Clinic at Toronto Western Hospital, University Health Network
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2027-02-12 (Estimated); Study Completion 2029-02-12 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory | For HC and TN > Neuropsychological assessments at baseline to screen for inclusion/exclusion criteria
  The Beck Depression Inventory (BDI) will be included in our battery of neuropsychological assessments that will be conducted on both HC and TN groups to screen for study inclusion and exclusion criteria. The BDI consists of 21 questions on which patients must score themselves on a scale from zero to three. The BDI is scored out of 63 with a score over 31 representing severe depression.
Behavioural Inhibition System | For HC and TN > Neuropsychological assessments at baseline to screen for inclusion/exclusion criteria
  The Behavioural Inhibition System (BIS) will be included in our battery of neuropsychological assessments that will be conducted on both HC and TN groups to screen for study inclusion and exclusion criteria. The BIS is a 20 question, self-assessment that measures trait sensitivity levels of the behavioral inhibition and activation systems.
Anxiety Sensitivity Index | For HC and TN > Neuropsychological assessments at baseline to screen for inclusion/exclusion criteria
  The Anxiety Sensitivity Index (ASI) will be included in our battery of neuropsychological assessments that will be conducted on both HC and TN groups to screen for study inclusion and exclusion criteria. The ASI is a six item scale that can outline different concerns someone could have regarding their anxiety.
Beck's Hopelessness Scale | For HC and TN > Neuropsychological assessments at baseline to screen for inclusion/exclusion criteria
  The Beck Hopelessness Scale (BHS) will be included in our battery of neuropsychological assessments that will be conducted on both HC and TN groups to screen for study inclusion and exclusion criteria.
Marlowe Crowne Scale | For HC and TN > Neuropsychological assessments at baseline to screen for inclusion/exclusion criteria
  The Marlowe Crowne Scale (MCS) will be included in our battery of neuropsychological assessments that will be conducted on both HC and TN groups to screen for study inclusion and exclusion criteria.
Childhood Trauma Questionnaire | For HC and TN > Neuropsychological assessments at baseline to screen for inclusion/exclusion criteria
  The Childhood Trauma Questionnaire (CTQ) will be included in our battery of neuropsychological assessments that will be conducted on both HC and TN groups to screen for study inclusion and exclusion criteria.
Structural magnetic resonance imaging (MRI) | For HC > MRI at baseline. For TN > MRI at baseline (pre-surgery) and at 6-month post-surgical)
  The investigators will acquire prospective longitudinal structural imaging data in 170 Trigeminal Neuralgia (TN) (pre-/6-months post-surgery) and 170 healthy controls (HC) and obtain topologies and volumes of the hippocampus (HPC) subfields using the brain imaging analysis software including HippUnfold and FreeSurfer. The investigators will also analyze amygdala (AMG) nuclei volumes using FreeSurfer. The group comparisons of the HPC and AMG will be done in both inter-group (TN vs. HC) and intra-group (pre- vs. post-surgery).
Mnemonic Similarity Test | For HC > MRI at baseline. For TN > MRI at baseline (pre-surgery) and at 6-month post-surgical)
  The Mnemonic Similarity Test will be used to compare HPC-dependent memory performance between TN and HC and examine the effect of surgery (pre- and post-) on performance. The investigators will assess whether HPC-dependent memory and HPC volumes/topologies normalize following surgical TN pain relief.
Fear of Pain Questionnaire III | For HC > pain-related fear and anxiety assessments at baseline. For TN >> pain-related fear and anxiety assessments at baseline (pre-surgery) and at 6-month post-surgical
  The Fear of Pain Questionnaire III (FPQ-III) will be used as one of the pain-related fear and anxiety assessments to assess pain-related fear and anxiety in TN and HC groups. The investigators will assess whether the abnormalities of the AMG nuclei volume will be normalized after surgery and will correlate these findings with validated pain-related fear and anxiety assessments. The FPQ-III is a 30 item assessment on which individuals rate how fearful they are of certain pain experiences on a scale from one to five.
Pain Catastrophizing Scale | For HC > pain-related fear and anxiety assessments at baseline. For TN >> pain-related fear and anxiety assessments at baseline (pre-surgery) and at 6-month post-surgical
  The Pain Catastrophizing Scale (PCS) will be used as one of the pain-related fear and anxiety assessments to assess pain-related fear and anxiety in TN and HC groups. The investigators will assess whether the abnormalities of the AMG nuclei volume will be normalized after surgery and will correlate these findings with validated pain-related fear and anxiety assessments. The PCS will help investigators quantify an individual's pain - how they feel and what they think about when experiencing something painful.
State-Trait Anxiety Inventory | For HC > pain-related fear and anxiety assessments at baseline. For TN >> pain-related fear and anxiety assessments at baseline (pre-surgery) and at 6-month post-surgical
  The State-Trait Anxiety Inventory (STAI) will be used as one of the pain-related fear and anxiety assessments to assess pain-related fear and anxiety in TN and HC groups. The investigators will assess whether the abnormalities of the AMG nuclei volume will be normalized after surgery and will correlate these findings with validated pain-related fear and anxiety assessments. The STAI is commonly used to measure trait and state anxiety. This assessment consists of 20 items for assessing trait anxiety and 20 for state anxiety, each of which are rated on a 4-point scale.
Pain Anxiety Symptoms Scale | For HC > pain-related fear and anxiety assessments at baseline. For TN >> pain-related fear and anxiety assessments at baseline (pre-surgery) and at 6-month post-surgical
  The Pain Anxiety Symptoms Scale (PASS-20) will be used as one of the pain-related fear and anxiety assessments to assess pain-related fear and anxiety in TN and HC groups. The investigators will assess whether the abnormalities of the AMG nuclei volume will be normalized after surgery and will correlate these findings with validated pain-related fear and anxiety assessments. The Pass-20 is a 20 item assessment that measures 4 distinct components of pain-related anxiety.
Functional Magnetic Resonance Imaging (fMRI) | For HC >ES task-fMRI at baseline. For TN >> ES task-based fMRI at baseline (pre-surgery) and 6-months post-surgery
  The experimental functional magnetic resonance imaging (fMRI) task that is specifically designed to measure episodic simulation (ES) using both neutral and pain-related cues will be conducted. ES measures the capacity to imagine specific future personal events and is heavily dependent on limbic integrity. This, along with the recalled pain memory interview will allow the investigators to correlate task-based fMRI findings with pain-recall discrepancies (discrepancies between recalled and initial pain ratings) and surgical response.
Recalled pain memory interview | For HC > recalled pain at baselines. For TN >> recalled pain at baseline (pre-surgery) and at 2 weeks and 6-month post-surgery
  The recalled pain interview, focused on the recall of pain events, will be conducted and analyzed with a specific focus on the discrepancies in pain recall (referred to as autobiographical memory, AM). Recalled Pain questionnaires will take place at baseline (~1 week prior to surgery, for the recall of pain onset and experience), acute recovery (2 weeks post-surgery) and 6 months post-surgery for recalled pain. These interview questionnaires will assess pain frequency, duration, intensity, fear, anxiety, unpleasantness, and interference.

SECONDARY OUTCOMES:
Structural Magnetic Resonance Imaging Cont. | For HC > MRI at baseline. For TN > MRI at baseline (pre-surgery) and at 6-month post-surgical)
  Group correlation between other AMG nuclei volumes and pain-related fear and anxiety questionnaires will be performed. The investigators will assess whether the abnormalities of other AMG nuclei volumes will be normalized after surgery and/or correlated with the validated pain-related fear and anxiety assessments.
The Rey Auditory Verbal Learning Test (RAVLT) | For HC > RAVLT at baseline. For TN > RAVLT at baseline (pre-surgery) and at 6-month post-surgical)
  Group correlation between other HPC subfield volumes and a second HPC-specific memory task using the Rey Auditory Verbal Learning Test (RAVLT) will be performed to evaluate multiple episodic memory functions in both inter-group (TN vs. HC) and intra-group (pre- vs. post-surgery).
Whole brain cortical-based analysis | For HC > MRI at baseline. For TN > MRI at baseline (pre-surgery) and at 6-month post-surgical)
  Group comparisons of other limbic structures will be performed, using the whole brain cortical-based analysis with a focus on the thickness of the anterior cingulate (ACC), insular, and medial prefrontal cortex (mPFC) cortices. The investigator will be focused on the dynamic changes of the cortical thickness in TN between i) TN vs. HC, and ii) pre- vs. post-surgical time points.
Impact of COVID-19 on pain population | For HC > COVID-19 related data at baseline. For TN > COVID-19 related data at baseline (pre-surgery) and at 6-month post-surgical)
  Medical and medication history including COVID-19-related experiences will be collected. The investigator will also address the biopsychological impacts of COVID-19 in our study cohort.
Sex- and gender-based analysis (SGBA) | For HC ad TN > SGBA at baseline as a part of the demographic data
  The investigator will target enrollment of a 50% male-to-female ratio. The investigator will also collect the gender identity data. SGBA will be conducted in all Aims and the distribution of gender data will determine whether we have sufficient power for detailed analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Mojgan Hodaie, MD, MSc, Principal Investigator — Department of Neurosurgery, Toronto Western Hospital, University Health Network
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Noorani A, Hung PS, Zhang JY, Sohng K, Laperriere N, Moayedi M, Hodaie M. Pain Relief Reverses Hippocampal Abnormalities in Trigeminal Neuralgia. J Pain. 2022 Jan;23(1):141-155. doi: 10.1016/j.jpain.2021.07.004. Epub 2021 Aug 8. PMID 34380093
- [Result] Hung PS, Noorani A, Zhang JY, Tohyama S, Laperriere N, Davis KD, Mikulis DJ, Rudzicz F, Hodaie M. Regional brain morphology predicts pain relief in trigeminal neuralgia. Neuroimage Clin. 2021;31:102706. doi: 10.1016/j.nicl.2021.102706. Epub 2021 May 25. PMID 34087549
- [Result] Vaculik MF, Noorani A, Hung PS, Hodaie M. Selective hippocampal subfield volume reductions in classic trigeminal neuralgia. Neuroimage Clin. 2019;23:101911. doi: 10.1016/j.nicl.2019.101911. Epub 2019 Jun 26. PMID 31491821
- [Result] Audrain S, McAndrews MP. Schemas provide a scaffold for neocortical integration of new memories over time. Nat Commun. 2022 Oct 2;13(1):5795. doi: 10.1038/s41467-022-33517-0. PMID 36184668
- [Result] Waisman A, Pavlova M, Noel M, Katz J. Painful reminders: Involvement of the autobiographical memory system in pediatric postsurgical pain and the transition to chronicity. Can J Pain. 2022 Jun 3;6(2):121-141. doi: 10.1080/24740527.2022.2058474. eCollection 2022. PMID 35692557
- [Result] Noel M, Rosenbloom B, Pavlova M, Campbell F, Isaac L, Page MG, Stinson J, Katz J. Remembering the pain of surgery 1 year later: a longitudinal examination of anxiety in children's pain memory development. Pain. 2019 Aug;160(8):1729-1739. doi: 10.1097/j.pain.0000000000001582. PMID 31335643
- See also: MedlinePlus related topics: Trigeminal Neuralgia — http://medlineplus.gov/trigeminalneuralgia.html
- See also: Genetic and Rare Disease Information Center Resources: Trigeminal Neuralgia — http://rarediseases.info.nih.gov/diseases/7805/trigeminal-neuralgia